CLINICAL TRIAL: NCT02185612
Title: EARN-Health: A Randomized Controlled Trial of the Effects of an Incentivized Savings Program on Depression, Anxiety, Substance Abuse, and Locus of Control
Brief Title: The EARN-Health Trial of Financial Savings and Health
Acronym: EARN-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 30641
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Depression; Anxiety; Alcohol Abuse; Tobacco Abuse
MeSH Terms: conditions — Depression; Anxiety Disorders; Alcoholism; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants will be randomized to a 1 year wait list. Participants take 0 month, 6 month, and 12 month surveys on depression, anxiety, alcohol and tobacco use, locus of control, and overall self-rated health.
- Savings program (Experimental): Participants will be randomized to the EARN.org online savings program for 6 months. Participants take 0 month, 6 month, and 12 month surveys on depression, anxiety, alcohol and tobacco use, locus of control, and overall self-rated health.
  Interventions: Behavioral: Savings program

INTERVENTIONS:
Behavioral: Savings program — The intervention is a web-based centralized savings account, which is a secure online account without fees. The account offers eligible savers nominal financial rewards for each deposit they make, as a financial incentive for savings.
  Arms: Savings program

SUMMARY:
The current literature in social epidemiology and public health suggests that low financial savings has an unsurprising negative relationship with subjective well-being, and increases the odds of making visits to a healthcare provider, receiving a chronic disease diagnosis, and experiencing medical disability. Earn.org is a community-based non-profit based in San Francisco with a mission to help low-income workers build lifelong savings habits and financial capability. The organization is one of the largest providers of "goal-based savings accounts" or "matched savings accounts" in the US. The investigators propose to conduct a randomized controlled trial to determine the health effects of Earn's savings program. Through this trial, the investigators will test three principal hypotheses: (1) Participants in the Earn account, as compared to a control group, are hypothesized to demonstrate improved scores on mental health scales assessing depression and anxiety.

(2) Participants in the Earn account, as compared to a control group, are hypothesized to experience lower odds of harmful behaviors associated with stress, specifically tobacco and alcohol abuse. The investigators hypothesize that the effect on behaviors will be of smaller effect size, and more delayed, than the effect on mental health outcomes, judging from similar effects observed in the micro-credit literature.

(3) The mediating variables between Earn account participation and beneficial health outcomes will include increased optimism and internal locus of control.

DETAILED DESCRIPTION:
The investigators plan to conduct an RCT comparing participants in the new EARN program against wait-listed control subjects. The program provides low-wage workers with incentives and rewards for savings. The program involves a web-based platform that permits eligible savers to create a centralized savings account, which is a secure online account without fees. The account offers eligible savers small monetary rewards for dollars saved each month. The investigators plan to conduct a baseline online month 0 survey and a follow-up 6 month and 12 month online survey among participants and wait-listed nonparticipants, with telephone follow-up to maximize 6- and 12-month survey completion. The surveys consist of previously-validated instruments to assess key health behaviors self-reported well-being, and require approximately 20 minutes each. The surveys includes the CDC Behavioral Risk Factor Surveillance System scales for assessing demographics and income, overall self-rated health, tobacco and alcohol use, depression and anxiety symptoms, and optimism and locus of control. Participants will receive prorated a gift card for each survey, to compensate participants for their time while avoiding a direct income effect of a cash incentive for participation.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking US residents
* ages 18 and older
* below 50% of the area median income
* have a regular Internet connection

Exclusion Criteria:

* non-English speakers
* non-US residents
* children,
* history of or current enrollment in other incentivized savings programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2016-10; Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Self-rated health scales | 12 months
  The following survey measures of self-rated health are taken from the validated CDC Behavioral Risk Factor Surveillance Study and will be recorded and reported from our study:
  H0) Would you say that in general your health, as compared to other people your age, is…?
  [ Excellent Very good Good Fair OR Poor ]
  H1) Please think about your physical health. This includes physical illness and injury. How many days during the past 30 days was your physical health not good?
  [Number from 0 to 30]
  H2) Now please think about your emotional health. This includes stress, depression, and anxiety. How many days during the past 30 days was your emotional health not good?
  [Number from 0 to 30]
  H3) During the past 30 days, for about how many days did poor physical or emotional health keep you from doing your usual activities, such as self-care, work, or recreation?
  [Number from 0 to 30]

SECONDARY OUTCOMES:
Depression and anxiety symptoms: yes/no questions | 12 months
  The following survey measures are taken from the validated Patient Health Questionnaire 8 and will be recorded and reported from our study:
  M1) Little interest or pleasure in doing things M2) Feeling down, depressed, or hopeless M3) Trouble falling asleep or staying asleep, or sleeping too much M4) Feeling tired or having little energy M5) Poor appetite or overeating M6) Feeling bad about yourself, or that you are a failure, or have let yourself or your family down M7) Trouble concentrating on things, such as reading the newspaper or watching television M8) Moving or speaking so slowly that other people could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual.
Alcohol abuse screening questions | 12 months
  The following survey measures of alcohol use are taken from the validated CDC Behavioral Risk Factor Surveillance Study and will be recorded and reported from our study:
  A1) During the past 30 days, how many days did you have at least one drink of any alcoholic beverage? This includes beer, wine, malt beverages, and liquor.
  Days in past 30 days
  A2) A drink of alcohol is 1 can or bottle of beer, 1 glass of wine, 1 can or bottle of wine cooler, 1 cocktail, or 1 shot of liquor. During the past 30 days, how many days per week or per month did you have at least one drink of any alcoholic beverage?
  A3) Considering all types of alcoholic beverages, how many times during the past 30 days did you have X [Script: X = 5 for men, X = 4 for women] or more drinks on an occasion?
Tobacco abuse screening questions | 12 months
  The following survey measures of tobacco use are taken from the validated CDC's Behavioral Risk Factor Surveillance Study and will be recorded and reported from our study:
  T0) Have you smoked at least 100 cigarettes in your entire life? yes no Script: If NO go to Part 5, else go to "T1"
  T1) Do you now smoke cigarettes every day, some days, or not at all? every day some days not at all
  T2) During the past 6 months, have you stopped smoking for one day or longer because you were trying to quit smoking?
Locus of control Likert scales | 12 months
  The following survey measures are taken from the validated Health and Retirement study to assess locus of control, and will be recorded and reported from our study::
  Please read the statements below and indicate the extent to which you agree with each statement. Select one of the following: Strongly Agree, Agree, Neutral, Disagree, or Strongly Disagree O1) In uncertain times, I expect the best O2) If something can go wrong for me, it will O3) I'm always optimistic about the future O4) I hardly ever expect things to go my way O5) I rarely count on good things happening to me O6) Overall, I expect more good things to happen to me than bad
Optimism Likert scales | 12 months
  The following survey measures are taken from the validated Health and Retirement study to assess optimism, and will be recorded and reported from our study::
  L1) I have little control over the things that happen to me L2) There is really no way I can solve some of the problems I have L3) There is little I can do to change many of the important things in my life L4) I often feel helpless in dealing with the problems of life L5) Sometimes I feel that I'm being pushed around in life L6) What happens to me in the future mostly depends on me L7) I can do just about anything I really set my mind to do
Spending behaviors | 12 months
  The following survey measures of spending behaviors will be recorded and reported from our study:
  S1) Over the past six months, would you say your household has been... Spending less money than you have had coming in. Spending more money than you have had coming in. Spending about the same amount of money that you have had coming in. S2) Over the past six months, which most accurately describes your household? We put aside money as savings every paycheck or every month. We put aside money as savings when we can, but not regularly. We didn't really put aside money as savings. S3) How much money did your household put aside as savings in an average month? We did not put aside savings in an average month. S4) Does your household have a monthly spending plan? Yes, and we mostly stick to it. Yes, but we don't really stick to it. No, we do not have a plan.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Basu, MD. PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basu S, Hamad R, White JS, Modrek S, Rehkopf DH, Cullen MR. The EARN-Health Trial: protocol for a randomised controlled trial to identify health effects of a financial savings programme among low-income US adults. BMJ Open. 2015 Oct 6;5(10):e009366. doi: 10.1136/bmjopen-2015-009366. PMID 26443663